CLINICAL TRIAL: NCT03481738
Title: Pyruvate Kinase Deficiency Global Longitudinal Registry
Acronym: PEAK Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AG348-C-008
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pyruvate Kinase Deficiency
Keywords: Glycolytic enzymopathy; Congenital Nonspherocytic hemolytic anemia (CNSA); PKD
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic, Congenital Nonspherocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PKD Diagnosed: Participants diagnosed with PK deficiency by the presence of 2 or more PKLR gene mutations as well as clinical features.

SUMMARY:
This study is an observational (ie, noninterventional), longitudinal, multicenter, global registry for patients with pyruvate kinase (PK) deficiency, a rare nonspherocytic hemolytic anemia.

This Registry will be open for enrollment for 7 years and all enrolled participants will be followed prospectively for a minimum of 2 years, and up to 9 years.

Data will be collected from participating Registry Physicians, participants, and, where appropriate, parents/guardians who have provided informed consent or assent (where relevant) and authorization pursuant to applicable laws and regulations.

Data should include demographic, clinical, and treatment data; and other data of relevance to the management of patients with PK deficiency. Annual chart review and data entry are expected in order to enhance longitudinal understanding of PK deficiency; however, no specific protocol schedule of assessment is required by this Registry protocol.

DETAILED DESCRIPTION:
Data will be submitted to the Registry via electronic case report forms (eCRFs). Relevant datasets, such as historical trial data, claims, medical records, or central lab data will be electronically integrated into the Registry or Registry reporting data sets.

Participants of all ages with a confirmed diagnosis of PK deficiency via genetic testing will be eligible to participate in this Registry. Diagnosis may be made on the basis of clinical features consistent with PK deficiency together with the presence of 2 or more PKLR gene mutations.

For novel or indeterminate PKLR gene mutations, participants will be deemed eligible if, in the opinion of the investigator, the reported PKLR gene mutations are sufficient to support a diagnosis of PK deficiency. Pyruvate kinase deficiency-relevant data will be entered by Registry Physicians or their designee for any and all participant visits. Disease parameters (eg, hemoglobin, reticulocyte counts), treatment and management options (splenectomy, transfusions, iron chelation, bone marrow transplant or pharmacological therapies) and resource utilization (eg, hospitalizations) will be evaluated to describe the natural history, treatments and outcomes, variability in clinical care and disease burden in patients with PK deficiency.

As a longitudinal observational study, the PK deficiency Registry may also serve as a data collection platform to address specific research objectives that may emerge over the duration of the study.

All data collection efforts will abide by this protocol and be prospectively disclosed in the Registry informed consent. If new assessments become of interest, they may be addressed via specific substudies (eg, patient-reported outcomes, biobanking), each requiring their own specific protocol and consent approved by Institutional Review Broad/Independent Ethics Committee (IRB/IEC). These studies may utilize a decentralized operational model with remote data capture. An IRB/IEC approved PEAK participant invitation process and participant self-opt-in registration may be utilized where country regulations and site policies allow.

This Registry, with the appropriate participant (and or parent/guardian) consent/assent, may incorporate retrospective data from other properly consented studies done for the purpose of examining the longitudinal natural history of PK deficiency. As necessary, data integration plan(s) will be developed to allow efficient and fit-for-purpose integration of data from other studies or data sets into this Registry.

Separate detailed statistical analysis plans (SAPs), addressing specific objectives, will be developed before the analyses during and at the end of the study. Due to the nature of the observational study, most statistical analyses will focus on descriptive statistics, including estimates and confidence intervals (CI) as appropriate. Additional statistical modeling of the data may be conducted. However, any p-values reported for hypothesis testing will be considered exploratory and therefore hypothesis-generating by nature. All data will be analyzed as collected in the database. Missing data, in general, will not be imputed; the modeling, eg, repeated measures mixed-effect models (MMRM) or generalized linear mixed effect model (GLIMMIX) will make use of all available data in the analyses. Any additional imputation techniques, if deemed necessary, will be discussed in the statistical analysis plan(s).

To ensure compliance with Good Clinical Practice and all applicable regulatory requirements, the Sponsor and its representatives will conduct and manage several plans that will ensure quality control. These will include:

* A documented sourcing procedure for all representatives and technology managing, collecting, or reporting on Registry data
* Assurance of FDA 21 CFR Part 11, EU-US Privacy Shield, and equivalent regulations regarding data security, controls, and audit trail of study data
* Assurance of the European Union regulation 2016/679 describing the appropriate use of personal data in scientific research
* Practices and methods for the protection of all participant privacy in relation to study data collection
* A training plan for site initiation and documentation
* Data entry guidelines that will assist all study sites with the completion of eCRFs
* A data monitoring and management plan that will outline the processes and procedures for reviewing, querying, and resolving data quality issues with study sites
* A site monitoring plan for the Sponsor and its representatives that will outline the frequency, requirements, and nature of the site monitoring visits for purposes of insuring data quality.

The Registry will be overseen by a Scientific Steering Committee, comprised of international experts involved in the research, diagnosis, and/or care of patients with PK deficiency. The Scientific Steering Committee's activities may include further defining the objectives and scientific direction of the Registry, advising on additional clinical data to be captured, and facilitating analysis and dissemination of Registry data via medical conferences and peer-reviewed publications.

ELIGIBILITY:
Inclusion Criteria:

* Participants of all ages with a confirmed diagnosis of PK deficiency via genetic testing are eligible to enroll;
* Participants will be considered for enrollment on the basis of clinical features consistent with PK deficiency together with the presence of 2 or more PKLR gene mutations. For novel or indeterminate PKLR gene mutations, participants will be deemed eligible if, in the opinion of the investigator, the reported PKLR gene mutations are sufficient to support a diagnosis of PK deficiency;
* The participant or the parent/guardian of the participant must be willing and able to give written informed consent and/or assent. E-consent or remote consent may be utilized where permissible as applicable if country regulations and site policies allow.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited or referred by physicians who treat hemolytic anemias at approximately 60 sites in approximately 20 countries.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Course of PK Deficiency | 9 years
  To develop an understanding of the longitudinal clinical implications of PK deficiency, including disease natural history, treatments and outcomes, and variability in clinical care and disease burden.

SECONDARY OUTCOMES:
Severity of Disease | 9 years
  To understand the prevalence, incidence, and severity of complications associated with PK deficiency.
Disease Impact on Pregnancy | 9 years
  To evaluate pregnancy outcomes.
Clinical Management Assistance | 9 years
  To provide a source of longitudinal data to assist physicians with clinical management of individual patients.
Global Repository | 9 years
  To act as a global repository for potential data from other properly consented PK deficiency-related studies to support aggregate and comparative analyses.

OTHER OUTCOMES:
Genetic | 9 years
  To examine a possible correlation between PKLR genotype and PK deficiency clinical phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Gallagher, VP, Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (52):
- United States (15):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
- Canada (3):
  - Saint Josephs Healthcare System, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - St. Justine Hospital, Montreal, Quebec
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Ustav hematologie a krevni transfuze, Prague
  - Fakultni nemocnice v Motole, Prague
- Copenhagen University Hospital, Herlev, Denmark
- Hopital Necker, Paris, France
- Germany (5):
  - Charite - Universitatsmedizin Berlin, Berlin
  - Evangelisches Krankenhaus Bielefeld gGmbH, Bielefeld
  - Universitatsklinikum Heidelberg, Heidelberg
  - Kinder- und Jugendarztpraxis, Munich
  - Universitatsklinikum Wurzburg, Würzburg
- St James's Hospital, Dublin, Ireland
- Italy (5):
  - Presidio Ospedaliero di Pescara, Pescara, Abruzzo
  - AOU dell'Universita degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - E O Ospedali Galliera, Genoa, Liguria
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale S Eugenio, Roma
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Portugal (3):
  - Centro Hospitalar E Universitario de Coimbra EPE, Coimbra
  - Centro Hospitalar Lisboa Central- Hospital Dona Estefania, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia / Espinho E.P.E, Porto
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, South Korea
- Spain (7):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Deu - PIN, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Tortosa Verge de la Cinta, Tortosa
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Siriraj Hospital Mahidol University, Bangkok, Thailand
- Hacettepe University Medical Faculty, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - Hammersmith Hospital, London, London, City of
  - Kings College Hospital, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grace RF, van Beers EJ, Vives Corrons JL, Glader B, Glenthoj A, Kanno H, Kuo KHM, Lander C, Layton DM, Pospisilova D, Viprakasit V, Li J, Yan Y, Boscoe AN, Bowden C, Bianchi P. The Pyruvate Kinase Deficiency Global Longitudinal (Peak) Registry: rationale and study design. BMJ Open. 2023 Mar 23;13(3):e063605. doi: 10.1136/bmjopen-2022-063605. PMID 36958777
- See also: Overview of the PEAK Registry — https://PEAKRegistry.com